CLINICAL TRIAL: NCT06829901
Title: The Effect of Entry Technique on Chorioamniotic Membrane Separation in Fetoscopic Laser Photocoagulation for Twin-To-Twin Transfusion Syndrome
Brief Title: The Effect of Uterine Entry In Fetoscopic Laser Photocoagulation for Twin-To-Twin Transfusion Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ahmed Nassr, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-56175
Record Dates: First submitted 2025-01-31; First posted 2025-02-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Twin to Twin Transfusion
Keywords: fetoscopic laser photocoagulation; TTTS; uterine entry; direct entry; Seldinger technique; chorioamniotic membrane separation; CAS
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Entry (Active Comparator): Surgeons will access the uterus to perform fetoscopic laser photocoagulation by inserting a sharp trocar through a small incision in the skin. The trocar is then removed and a small tube called a cannula is left in place.
  Interventions: Procedure: Fetoscopic Laser Photocoagulation
- Seldinger Technique (Active Comparator): Surgeons will access the uterus to perform fetoscopic laser photocoagulation by inserting needle through a small incision in the skin and running a guide wire through the needle so a thin tube called a cannula can be placed over the wire.
  Interventions: Procedure: Fetoscopic Laser Photocoagulation

INTERVENTIONS:
Procedure: Fetoscopic Laser Photocoagulation — Patients who choose to undergo fetoscopic selective laser photocoagulation for complicated monochorionic-diamniotic twin pregnancies with twin-to-twin transfusion syndrome will be offered participation in the study. All participants will undergo selective laser photocoagulation and entry into the uterus will be achieved using one of two accepted methods, either direct entry or the Seldinger technique.

SUMMARY:
The purpose of this study is to evaluate whether the entry technique surgeons use to get inside the uterus to perform fetoscopic laser photocoagulation for twin-to-twin transfusion syndrome has an effect on the rates of chorioamniotic membrane separation.

DETAILED DESCRIPTION:
Patients who choose to undergo fetoscopic selective laser photocoagulation (SFLP) at Texas Children's Fetal Center will be offered participation in this research study by study investigators. Description of study rationale and design and a focused interview by the study coordinator to afford potential participants a formal opportunity to examine what they have learned about the research study in the course of their evaluation and discuss how they feel about enrolling in the research study. Once the patient is deemed eligible the informed consent process will be reviewed. If patients elect to participate in the study, informed consent will be obtained, and participants will be provided a copy of the signed consent.

After consent has been obtained, participants will be randomized into two groups ("direct entry" and "Seldinger technique").

Procedure: Selective laser photocoagulation (SFLP) is standard of care for the treatment of complicated monochorionic twin pregnancies. Entry into the uterus for SFLP is achieved under ultrasound guidance using one of two accepted methods, direct entry or the Seldinger technique. Intravenous sedation with local anesthesia at the site of insertion has been found to provide sufficient maternal anesthesia for the procedure.

Group I - Direct entry: The surgeon will gain access to the uterus by inserting a sharp trocar through a small incision in the skin. After access has been established, the trocar is removed and a small tube called a cannula is left in place.

Group II - Seldinger technique: The surgeon will gain access to the uterus by inserting needle through a small incision in the skin and run a guide wire through the needle so a thin tube called a cannula can be placed over the wire.

Follow-Up:

Participants will be monitored after the procedure and upon discharge from the hospital they are free to resume care with their primary doctor. Investigators will collect follow-up data on the health of the participant and the babies until the babies turn one month old.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and elect to undergo fetoscopic selective laser photocoagulation for complicated monochorionic-diamniotic twin pregnancies with twin-to-twin transfusion syndrome.

Exclusion Criteria:

* Patients who do not elect to undergo fetoscopic laser photocoagulation for the treatment of complicated monochorionic-diamniotic twin pregnancies with twin-to-twin transfusion syndrome.
* Triplets and higher order multiple gestations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Immediate Chorioamniotic Membrane Separation (CAS) | Up to hospital discharge post-procedure (up to 5 days)
  Number of participants that have chorioamniotic membrane separation within 24 hours of the procedure.

SECONDARY OUTCOMES:
Rate of Chorioamniotic Membrane Separation (CAS) | From the post-surgical period (outside the first 24 hours) until delivery, up to 25 weeks
  Number of participants that have chorioamniotic membrane separation outside the first 24 hours hours following the procedure
Gestational Age at Delivery | At delivery
  Gestational age at the time of delivery
Preterm Birth | At delivery
  Number of participants that deliver at <37 weeks gestation
Procedure to Delivery Interval | At delivery
  Days between the participant's procedure and when the babies are delivered
Placental Abruption | Up to hospital discharge post-procedure (up to 5 days)
  As measured by presence in medical record
Chorioamnionitis | Up to hospital discharge post-procedure (up to 5 days)
  As measured by presence in medical record
Septostomy | Up to hospital discharge post-procedure (up to 5 days)
  As measured by presence in medical record
Preterm Premature Rupture of Membranes (PPROM) | At delivery
  As measured by presence in medical record

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nassr, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital - Pavilion for Women, Houston, Texas, United States